CLINICAL TRIAL: NCT04057222
Title: Effect of Need to Void on Rectal Sensory Function in Multiple Sclerosis, a Manometric Study
Brief Title: Effect of Need to Void on Rectal Sensory Function in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gérard Amarenco (Other)
Responsible Party: Sponsor-Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon Hospital, Pierre and Marie Curie University
Organization: Pierre and Marie Curie University (Other)
Other Study IDs: GRC-01GREEN
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis; Anorectal Disorders; Bladder Dysfunction
Keywords: Rectal sensory function; Multiple sclerosis; anorectal disorders; Fecal incontinence; constipation; bladder sensation
MeSH Terms: conditions — Multiple Sclerosis; Rectal Diseases; Fecal Incontinence; Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients included: Patient with multiple sclerosis and anorectal symptoms, with indication to realize a anorectal manometry, age > 18
  A first record of rectal sensory function will be at strong desire to void. A second record will be after void. Rectal sensory function records consist on an anorectal manometry with 3 measures of external anal sphincter resting pressure, 5 measures of RAIR, 1 measure of perception, constant sensation to need to defecate and maximum tolerable threshold volumes.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Only propose water and wait for need to void

SUMMARY:
Multiple sclerosis causes demyelinating lesions, which can induce multiple symptoms. Ano-rectal avec urinary disorders are frequent due to specific lesions in inhibitor/activator encephalic centers, or interruption on medullary conduction. It seems to be evident that anorectal and urinary disorders are link, because of similar anatomic ways and control process.

To our knowledge several studies test the effect of rectal distension and bladder sensory function but only one study examined the effect of bladder filling on rectal sensitivity on healthy people. The effect of bladder filling on rectal sensory function in patient with neurological disease stay unknown, while dysfunction often occur concomitant, and therapeutic actions in one organ may influence function of the other.

Anorectal manometry is the gold standard for the evaluation of rectal sensory function and the volume of constant sensation to need to defecate is reported in literature as the most reproducible measure.

Primary aim is to assess the effect of need to void on volume of constant sensation to need to defecate in multiple sclerosis with anorectal symptoms. Secondary aim is to identify the effect of need to void on modulation of rectoanal inhibitory reflex (RAIR) and external anal sphincter resting pressure.

Patient with multiple sclerosis over 18 years old, consulting for anorectal disorders in a tertiary center, with an indication to realize an anorectal manometry are included.

History and treatment, height, weight, Expanded Disability Status Scale (EDSS), anorectal and urinary symptoms severity by Bristol, Neurogenic Bowel Dysfunction (NBD), Cleveland, Kess, Urinary Symptom Score (USP) scores, and last urodynamic data are recorded. Patient are asked to drink water until they feel a strong need to void, for which they would go to urinate at home. 3 void volume with portable sonography are done, and the higher is recorded.

Anorectal manometries are realized by the same doctor, in a specific place, with calm. Before the manometric examination, thermal and vibratory sensory thresholds on the right hand are collected. The patient is then placed in a left lateral position. Then the anorectal manometry's catheter is inserted and collect of the external anal sphincter resting pressure begins. Then the investigator proceed to search for RAIR by 5 brief distensions of the intrarectal balloon with increasing volumes of 10 mL from 10 mL to 50 mL. Finally, the investigator collect the threshold volumes of perception, need and maximum tolerable by gradually distending the intra-rectal balloon to 5 mL/s from 0 mL to 300 mL. Toilets are just next to the table of examination.

Next, patient can urinate. 3 post void residual volume with portable sonography are done, and the higher is recorded.

The same tests are realized after urinate, in the same order. After the classical complete manometry was performed.

Primary outcome is the volume of constant sensation to need to defecate Secondary outcomes are the modulation of RAIR and the external anal sphincter resting pressure. Manometric data are collected.

Influence of age, EDSS, severity of symptoms, manometric data and detrusor overactivity on rectal sensory function will be study in secondary analysis.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis
* > 18 years old
* Anorectal disorders

Exclusion Criteria:

* full rectal ampullae
* No bladder sensation
* inability to understand simple orders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with multiple sclerosis over 18 years old, consulting for anorectal disorders in a tertiary center, with an indication to realize an anorectal manometry are included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-07-26 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
Variation of volume of rectal constant sensation to need to defecate | 1 Day
  Difference between volume of rectal constant sensation to need to defecate at strong desire to void and post void, collected by patient declaration when distending the intra-rectal balloon by manual air insufflation at 5 mL/s during

SECONDARY OUTCOMES:
Variation of amplitude modulation of the RAIR between strong desire to void and just after | 1 Day
  Difference between amplitude modulation of the RAIR at strong desire to void and post void calculated by difference between two non-successive residual pressure values on five successive distension volumes.
Variation of duration modulation of the RAIR between strong desire to void and just after | 1 Day
  Difference between duration modulation of the RAIR at strong desire to void and post void calculated by difference between two non-successive residual pressure values on five successive distension volumes.
Variation of external anal sphincter resting pressure between strong desire to void and just after | 1 Day
  Difference between external anal sphincter resting pressure at strong desire to void and post void

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PUPH, Principal Investigator — Sorbonne Université, GRC 001, GREEN, AP-HP, Hôpital Tenon, Paris, France
Locations (1):
- department of Neuro-Urology, Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pouyau C, Grasland M, Leroux C, Chesnel C, Turmel N, Sheikh Ismael S, Le Breton F, Amarenco G, Hentzen C. Relationship between desire to void and bladder capacity and rectal sensory function in patients with multiple sclerosis and anorectal disorders. Neurourol Urodyn. 2020 Apr;39(4):1129-1136. doi: 10.1002/nau.24330. Epub 2020 Mar 12. PMID 32163639